CLINICAL TRIAL: NCT06305065
Title: Open and Closed Platform Robotic-assisted Versus Conventional Total Knee Arthroplasty: a Randomised Controlled Trial
Brief Title: Open and Closed Platform Robotic-assisted Versus Conventional Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024.089
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
Keywords: Knee Osteoarthritis; Knee OA; Total Knee Arthroplasty; Robotic-assisted TKA procedure
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: Subjects will be randomly assigned to the KUNWU navigational or CORI Surgical System or conventional manual instrumentation groups according to a balanced randomization procedure using a 1:1:1 allocation ratio. To ensure balanced group assignment, a block randomization schedule will be generated. All subjects who sign the ICF and meet all inclusion and exclusion criteria will be randomized in a 1:1:1 randomization allocation ratio. The block size should be sufficiently small to allow approximately equal allocation of subjects in each group should the study be terminated prematurely whilst also being large enough so as the next treatment cannot be guessed. The study is non-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KUNWU Navigation TKA procedure (Experimental): Yuanhua Orthopaedic Robotic Systems, KUNWU, is an open-platform robotic system that does not restrict surgeons in choosing the type of prosthesis implant. It is the only Orthopaedic Robotic System in Hong Kong registered with the HK Department of Health Medical Devices Control Office (MDCO) as an open platform system. Unlike other manufacturer's implant-based robots (closed systems), Yuanhua's objective is to provide maximum flexibility in choosing the best implant for each patient. Closed system robots not only impact the surgeon's choice of implant for an individual patient but also affect the hospital's implant purchases over multiple years without any negotiation power on pricing. This business model is often referred to as a "razor and razor blade" model.
  Interventions: Procedure: KUNWU Navigation TKA procedure
- CORI Surgical System TKA procedure (Experimental): REAL INTELLIGENCE™ CORI™ (CORI Surgical System) is a computer-assisted orthopedic surgical system. CORI Surgical System is designed to aid surgeons in planning and executing a procedure involving bone preparation for total knee arthroplasty (TKA) procedures.
  CORI Surgical System is comprised of a console control unit, optical tracking camera, primary and secondary input displays (tablet and optional display monitor), and foot pedal. The CORI Surgical System software consists of a patient and user management module, a surgical planner, and an intra-operative cutting module.
  Interventions: Procedure: CORI Surgical System TKA procedure
- Conventional TKA procedure (Active Comparator): This group will perform the standard TKA procedure.
  Interventions: Procedure: Conventional TKA procedure

INTERVENTIONS:
Procedure: KUNWU Navigation TKA procedure — In terms of technical specifications, KUNWU is the only robotic arm with seven degrees of freedom, while other systems have a maximum of six. The ergonomic and user-friendly design of the system contributes to physical relief and simplified instrument handling, which enhances surgical precision and reduces cognitive stress.
  KUNWU's navigation system boasts a refresh rate of 335Hz, which is significantly higher than the current 60Hz rate of other navigation systems. This high refresh rate provides a clear and visually captivating display of the navigation procedure, eliminating blurriness and indecipherable output. It enables surgeons to react promptly during live procedures, enhancing safety for both clinicians and patients and reducing potential complications and hospitalization.
  Arms: KUNWU Navigation TKA procedure
Procedure: CORI Surgical System TKA procedure — The CORI Surgical System (Smith and Nephew®) represents one of such recent advances in robotics that it can assist surgical planning, and increase the accuracy of implant position due to real-time feedback during the procedure (bone resection, implant position, ligamentous balance).
  Arms: CORI Surgical System TKA procedure
Procedure: Conventional TKA procedure — Total knee arthroplasty (TKA) is a highly successful and frequently performed surgical treatment to reduce disability caused by end-stage osteoarthritis and other conditions affecting articular cartilage. Technical outcomes for TKA are excellent, with favorable postoperative health-related quality of life. Also, survivorship of primary knee replacements is excellent with reported survivorship of 82.3% at 25 years. TKA has traditionally been indicated in the elderly population with relatively sedentary lifestyles, but more active, younger patients (<55) are receiving TKA due to the desire for a pain-free, active lifestyle with the demand projected to continue to increase for this group. A recent systematic review has shown that functional outcomes are similar in this population compared to elderly patients with no increase in the burden of revision.
  Arms: Conventional TKA procedure

SUMMARY:
REAL INTELLIGENCE™ CORI™ (CORI Surgical System) is a computer-assisted orthopedic surgical system. CORI Surgical System is designed to aid surgeons in planning and executing a procedure involving bone preparation for total knee arthroplasty (TKA) procedures.

CORI Surgical System is comprised of a console control unit, optical tracking camera, primary and secondary input displays (tablet and optional display monitor), and foot pedal. The CORI Surgical System software consists of a patient and user management module, a surgical planner, and an intra-operative cutting module.

Yuanhua Orthopaedic Robotic Systems, KUNWU, is an open-platform robotic system that does not restrict surgeons in choosing the type of prosthesis implant. It is the only Orthopaedic Robotic System in Hong Kong registered with the HK Department of Health Medical Devices Control Office (MDCO) as an open platform system. Unlike other manufacturer's implant-based robots (closed systems), Yuanhua's objective is to provide maximum flexibility in choosing the best implant for each patient. Closed system robots not only impact the surgeon's choice of implant for an individual patient but also affect the hospital's implant purchases over multiple years without any negotiation power on pricing. This business model is often referred to as a "razor and razor blade" model.

The primary objective of this study is to evaluate the use of open and closed platform robotic-assisted TKA procedure in achieving post-operative leg alignment as compared to procedures using standard instruments. The secondary objective of this study is to assess the safety and performance of the robotic-assisted TKA procedure up to 12 months after surgery as compared to procedures using conventional manual instruments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a suitable candidate for a robotic-assisted TKA procedure
2. Subject requires a cemented TKA as a primary indication that meets any of the following condition:

   * Degenerative joint disease, including osteoarthritis
   * Rheumatoid arthritis
   * Avascular necrosis
   * Requires correction of functional deformity
   * Requires treatment of fractures that were unmanageable using other techniques
3. Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery)
4. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethical Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
5. Subject plans to be available through two (2) year postoperative follow-up.
6. Applicable routine radiographic assessment is possible.

Exclusion Criteria:

1. Subject requires a TKA on the index joint as a revision for a previously failed surgery, or has the need for complex implants, or any other implant than a standard TKA (e.g. stems, augments, or custom made devices).
2. Subject has been diagnosed with post-traumatic arthritis.
3. Subject requires bilateral TKA.
4. Subject does not understand the language used in the Informed Consent Form.
5. Subject does not meet the indication or is contraindicated for TKA according to the specific Smith+Nephew Knee System's Instructions For Use (IFU).
6. Subject has active infection or sepsis (treated or untreated).
7. Subject is morbidly obese with a body mass index (BMI) greater than 40.
8. Subject is pregnant or breast feeding at the time of surgery.
9. Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
10. Subject has a condition(s) that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
11. Subject in the opinion of the Investigator has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.
12. Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative leg alignment - Hip-knee-ankle axis (HKA axis) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The primary objective of this study is to evaluate the use of open and closed platform robot in TKA procedure in achieving post-operative leg alignment as compared to procedures using conventional manual instruments.
  The mechanical axis of the lower limb is calculated as the angle between the following two lines: the first line drawn from the centre of the femoral head to the centre of the knee joint, and the second line is drawn from the centre of the knee to the centre of the ankle joint.
  Record the correct angle in degrees for 'Leg Alignment on Standing long leg X-Ray - Provide angle and select one position Angle (neutral/ varus/ valgus)'. The angular deviation will be measured from the neutral position (180°).

SECONDARY OUTCOMES:
Lateral View | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  Femoral Flexion Angle: The lateral view femoral flexion angle (X) is obtained from the intersection of a line from the center of the femoral implant to the top of the femur with a line through the femoral canal. The angle is measured on the proximal side of the intersection Tibial Lateral Angle: The lateral view tibial angle (Y) is the angle obtained from the intersection of a line drawn parallel to the bottom of the tibial base insert and a line through the center of the tibial base and the tibial canal.
Standard Radiographic Evaluation - Femoral coronal alignment (FCA) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The femoral prosthesis coronal alignment is the degree to which the femoral prosthesis is deviated from the mechanical axis of the lower extremity.
Standard Radiographic Evaluation - Femoral sagittal alignment (FSA) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The femoral sagittal alignment gives the flexion of the femoral component in lateral view. The flexion of the component is the angle formed between the mechanical axis of the femur in the sagittal plane and the line perpendicular to the tangent of the distal portion of the femoral component.
Standard Radiographic Evaluation - Femoral component rotation (FCR) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The rotation of the femoral component is defined on the axial section of the post-operative CT scan. The angle of deviation between the radiographic trans-epicondylar axis (rTEA) and femoral prosthesis posterior condylar line (FPPCL) is the amount of femoral component rotation.
Standard Radiographic Evaluation - Tibial coronal alignment (TCA) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The tibial prosthesis coronal alignment gives the varus/valgus angulation of the prosthesis which affects the mechanical axis of the lower limb.
Standard Radiographic Evaluation - Tibial slope | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The tibial slope is calculated pre-operatively as the angle between the perpendicular to the anatomical axis of the tibia and the line joining the anterior and posterior point of the tibial surface on the lateral view.
Standard Radiographic Evaluation - Joint line distance | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  In this study, the tip of the fibular head is used as the fixed bony point to calculate the joint line pre- and post-operatively. Pre-operatively, the perpendicular distance from the tip of the fibular head to the joint line of knee was termed as the joint line distance. Post-operatively, the perpendicular distance from the tip of the fibular head to the line joining the medial and lateral femoral prosthesis was termed as the joint line distance.
Knee Society Score (KSS) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component. The KSS consists of 34 questions and provides sub-scores across 4 dimensions, including Objective Knee Score, Symptoms, Subject Satisfaction Score, Subject Expectation, and Functional Knee Score.
  The Objective Knee Score is rated by the clinician and assesses a range of clinical outcomes: TKA alignment, stability, range of motion (ROM) and symptoms.
  The KSS is an instrument assessing patient's pain and functionality based on a series of questions interviewed by a clinician. The validated questionnaire combines the objective physician derived component with a subjective patient derived component which evaluates pain, functionality, satisfaction and fulfillment of expectations. The results will be calculating the total score with 100 being the highest and 0 the lowest.
Oxford Knee Score (OKS) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The OKS will be collected at the pre-operative visit and 6 weeks, 6 months, and 12 months after surgery.
  The OKS is a Patient Reported Outcome (PRO) questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty. The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome. The benefit to this questionnaire is that it is short, practical, reliable, valid and sensitive to clinically important changes over time.
  A paper questionnaire will be provided by the Sponsor to be completed by the subject. Responses for the OKS will then be recorded.
HEALTH ECONOMICS/QUALITY OF LIFE - EQ-5D-5L | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system is used to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas.
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health)
Forgotten Joint Score (FJS) | pre-operative visit, day of surgery, 6 weeks, 6 months, and 12 months after surgery
  The FJS will be collected at 6 weeks, 6 months, and 12 months after surgery. A paper questionnaire will be provided to be completed by the subject.
  The FJS comprises measures for the assessment of joint-specific patient reported outcomes. This questionnaire focuses on the study subject's awareness of the partially or fully replaced knee joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. Subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.
  A paper questionnaire will be provided to be completed by the subject. Responses for the FJS will then be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers